CLINICAL TRIAL: NCT06073613
Title: Periodontal Status in Patients With Chronic Skin Diseases: a Pilot Study
Brief Title: Periodontal Status in Patients With Chronic Skin Diseases
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Hoa Ho Thi, Inverstigator, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: HoChiMinhCityUMP_FOS
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Periodontal Diseases; Psoriasis; Atopic Dermatitis; Autoimmune Bullous Dermatosis; Systemic Lupus Erythematosus
Keywords: chronic skin disease; periodontal status; oral lesions
MeSH Terms: conditions — Periodontal Diseases; Psoriasis; Dermatitis, Atopic; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: healthy individuals, aged 18 years or older and free of chronic skin diseases, willing to participate in the study
  Interventions: Diagnostic Test: oral health status
- Patients with CSDs: Patients with CSDs (psoriasis, atopic dermatitis, autoimmune bullous diseases, or systemic lupus erythematosus,…) were diagnosed by the dermatologists with over 5 years of experience and supportive laboratory tests, aged 18 years or older, and willing to participate in the study
  Interventions: Diagnostic Test: oral health status

INTERVENTIONS:
Diagnostic Test: oral health status — * CSDs medical records: Information related to epidemiological characteristics and chronic inflammatory skin conditions (psoriasis, atopic dermatitis, autoimmune bullous diseases, or systemic lupus erythematosus,…) were recorded from medical records:
    * Pemphigus
    * Mixed connective tissue disease
    * Atopic dermatitis
    * Psoriasis
    * Erythroderma
  * oral health status: oral clinical parameters were evaluated:
    * Full mouth bleeding on probing scores
    * Pocket probing depth
    * Clinical attachment level
    * debris index
    * calculus index
    * the number of oral lesions
  Other Names: CSDs medical records

SUMMARY:
Objective: This study aimed to evaluate and compare the periodontal status of chronic skin disease (CSD) patients with healthy controls.

Material and method: 109 patients and 37 healthy subjects were included in this study. Parameters evaluated included bleeding on probing index (BOP), periodontal pocket depths (PPD), clinical attachment level (CAL), simplified debris index (DI), simplified calculus index (CI), and the presence of oral lesions. Clinical parameters were measured and compared in the two groups. The significant level was set at 0.05.

DETAILED DESCRIPTION:
Patients with CSDs (psoriasis, atopic dermatitis, autoimmune bullous diseases, or systemic lupus erythematosus,…) were diagnosed by the dermatologists with over 5 years of experience and supportive laboratory tests, aged 18 years or older, and willing to participate in the study. The control group included healthy individuals, aged 18 years or older and free of chronic skin diseases. These individuals were willing to participate in the study and would be used as a comparison group for the case group.

Clinical parameter collection Information related to epidemiological characteristics and chronic inflammatory skin conditions were recorded from medical records and oral health status was collected from clinical examination conducted by postgraduate doctors and lecturers of the Faculty of Odonto-Stomatology, University of Medicine and Pharmacy at Ho Chi Minh City. The investigators were trained by a specialist in public dentistry and had intra-rater and inter-rater reliability of more than or equal to 0.8.

The following oral clinical parameters were evaluated:

1. Full mouth bleeding on probing scores (BOP): BOP was recorded and considered positive when bleeding occurred within 20 seconds after the probe was removed after application with light pressure. A bleeding percentage was calculated for each patient by dividing the total number of positive bleeding sites by the total number of probed sites.
2. Pocket probing depth (PPD) was measured from the gingival margin to the base of the gingival sulcus/ periodontal pocket with the aid of a University of North Carolina (UNC) 15-mm periodontal probe.
3. Clinical attachment level (CAL) was measured from the cemento-enamel junction (CEJ) to the base of the gingival sulcus/ periodontal pocket with the aid of a UNC periodontal probe. The CAL was considered zero if the attachment was at the level of the CEJ. If the free gingival margin was coronal to the CEJ, the CAL was determined by measuring the PPD and subtracting the distance from the CEJ to the free gingival margin. When the free gingival margin was apical to the CEJ, the CAL was determined by measuring the distance from the CEJ to the free gingival margin and adding it to the PPD.
4. debris index (DI), and (5) calculus index (CI), which were evaluated pertaining to the Simplified Oral Hygiene Index (OHI-S) as suggested by Green and Vermillion (1964)

(6) the number of oral lesions. Probed sites were classified into three different categories of PPD and CAL (≤ 3 mm, 4-5 mm, > 6mm).

The investigator examined one tooth (index teeth) from each sextant, including the incisor, left and right molar regions for both the maxillary and mandibular dental arches, to record the CAL, DI, and CI.

Statistics analysis All statistical analysis was performed using Jeffrey's Amazing Statistics Program (JASP) software, version 0.17.2.1 (University of Amsterdam, Amsterdam, The Netherlands). The normality of distribution of the data was verified using the Shapiro-Wilk test. For variables that were under normal distribution, independent t-test test was used for detecting the statistically significant differences among two groups. For variables that were not normally distributed, Mann-Whitney test was used to compare among two groups. P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient CSDs:

  * were diagnosed in CSDs (psoriasis, atopic dermatitis, autoimmune bullous diseases, or systemic lupus erythematosus...) by the dermatologists with over 5 years of experience and supportive laboratory tests
  * aged 18 years or older
  * willing to participate in the study
* Control group:

  * aged 18 years or older
  * free of chronic skin diseases

Exclusion Criteria:

* Toothless
* Limited mouth opening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A prospective case-control study was conducted at Ho Chi Minh City Hospital of Dermato-Venereology in February 2023 to assess the periodontal status of patients with CSDs. The study included 109 patients with CSDs, including psoriasis, atopic dermatitis, lupus, and common autoimmune bullous skin diseases, and 37 healthy controls.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Full mouth bleeding on probing scores (BOP) | baseline
  BOP was recorded and considered positive when bleeding occurred within 20 seconds after the probe was removed after application with light pressure. A bleeding percentage was calculated for each patient by dividing the total number of positive bleeding sites by the total number of probed sites
Pocket probing depth (PPD) | baseline
  PPD was measured from the gingival margin to the base of the gingival sulcus/ periodontal pocket with the aid of a University of North Carolina (UNC) 15-mm periodontal probe
Clinical attachment level (CAL) | Baseline
  was measured from the cemento-enamel junction (CEJ) to the base of the gingival sulcus/ periodontal pocket with the aid of a UNC periodontal probe. The CAL was considered zero if the attachment was at the level of the CEJ. If the free gingival margin was coronal to the CEJ, the CAL was determined by measuring the PPD and subtracting the distance from the CEJ to the free gingival margin. When the free gingival margin was apical to the CEJ, the CAL was determined by measuring the distance from the CEJ to the free gingival margin and adding it to the PPD
debris index (DI) | Baseline
  DI were evaluated pertaining to the Simplified Oral Hygiene Index (OHI-S) as suggested by Green and Vermillion (1964)
calculus index (CI) | Baseline
  CI were evaluated pertaining to the Simplified Oral Hygiene Index (OHI-S) as suggested by Green and Vermillion (1964)
the number of oral lesions | Baseline
  Probed sites were classified into three different categories of PPD and CAL (≤ 3 mm, 4-5 mm, > 6mm)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Trong Nguyen, PhD, Study Director — Ho Chi Minh City Hospital of Dermato-Venereology, Ho Chi Minh City, Vietnam; Thuy Thu Nguyen, PhD, Study Director — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh city, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
Study conception and design by groups of 8 researchers working at Ho Chi Minh City Hospital of Dermato-Venereology, Ho Chi Minh City, Vietnam and Faculty of Odonto-stomatology, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Arduino PG, Farci V, D'Aiuto F, Carcieri P, Carbone M, Tanteri C, Gardino N, Gandolfo S, Carrozzo M, Broccoletti R. Periodontal status in oral mucous membrane pemphigoid: initial results of a case-control study. Oral Dis. 2011 Jan;17(1):90-4. doi: 10.1111/j.1601-0825.2010.01709.x. PMID 20659265
- [Background] Lo Russo L, Gallo C, Pellegrino G, Lo Muzio L, Pizzo G, Campisi G, Di Fede O. Periodontal clinical and microbiological data in desquamative gingivitis patients. Clin Oral Investig. 2014 Apr;18(3):917-25. doi: 10.1007/s00784-013-1038-8. Epub 2013 Jul 31. PMID 23900791
- [Background] Lo Russo L, Guiglia R, Pizzo G, Fierro G, Ciavarella D, Lo Muzio L, Campisi G. Effect of desquamative gingivitis on periodontal status: a pilot study. Oral Dis. 2010 Jan;16(1):102-7. doi: 10.1111/j.1601-0825.2009.01617.x. Epub 2009 Sep 4. PMID 19735453
- [Background] Ramon-Fluixa C, Bagan-Sebastian J, Milian-Masanet M, Scully C. Periodontal status in patients with oral lichen planus: a study of 90 cases. Oral Dis. 1999 Oct;5(4):303-6. doi: 10.1111/j.1601-0825.1999.tb00094.x. PMID 10561718
- [Background] Schellinck AE, Rees TD, Plemons JM, Kessler HP, Rivera-Hidalgo F, Solomon ES. A comparison of the periodontal status in patients with mucous membrane pemphigoid: a 5-year follow-up. J Periodontol. 2009 Nov;80(11):1765-73. doi: 10.1902/jop.2009.090244. PMID 19905946
- [Background] Thorat MS, Raju A, Pradeep AR. Pemphigus vulgaris: effects on periodontal health. J Oral Sci. 2010 Sep;52(3):449-54. doi: 10.2334/josnusd.52.449. PMID 20881339
- [Background] Tricamo MB, Rees TD, Hallmon WW, Wright JM, Cueva MA, Plemons JM. Periodontal status in patients with gingival mucous membrane pemphigoid. J Periodontol. 2006 Mar;77(3):398-405. doi: 10.1902/jop.2006.050113. PMID 16512754
- [Background] Jascholt I, Lai O, Zillikens D, Kasperkiewicz M. Periodontitis in oral pemphigus and pemphigoid: A systematic review of published studies. J Am Acad Dermatol. 2017 May;76(5):975-978.e3. doi: 10.1016/j.jaad.2016.10.028. Epub 2016 Dec 28. PMID 28038889
- [Background] Macklis P, Adams K, Kaffenberger J, Kumar P, Krispinsky A, Kaffenberger B. The Association Between Oral Health and Skin Disease. J Clin Aesthet Dermatol. 2020 Jun;13(6):48-53. Epub 2020 Jun 1. PMID 32884621
- [Background] Rai NP, Kumar P, Mustafa SM, Divakar DD, Kheraif AA, Ramakrishnaiah R, Vellapally S, Dalati MH, Parine NR, Anil S. Relation Between Periodontal Status and Pre-Cancerous Condition (Oral Lichen Planus): A Pilot Study. Adv Clin Exp Med. 2016 Jul-Aug;25(4):763-6. doi: 10.17219/acem/59014. PMID 27629852
- [Background] Listgarten MA. Pathogenesis of periodontitis. J Clin Periodontol. 1986 May;13(5):418-30. doi: 10.1111/j.1600-051x.1986.tb01485.x. PMID 3522650
- [Background] Offenbacher S, Heasman PA, Collins JG. Modulation of Host PGE2 Secretion as a Determinant of Periodontal Disease Expression. J Periodontol. 1993 May;64 Suppl 5S:432-444. doi: 10.1902/jop.1993.64.5s.432. PMID 29539680
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Result] Akman A, Kacaroglu H, Yilmaz E, Alpsoy E. Periodontal status in patients with pemphigus vulgaris. Oral Dis. 2008 Oct;14(7):640-3. doi: 10.1111/j.1601-0825.2008.01445.x. PMID 18627505